CLINICAL TRIAL: NCT02781584
Title: A Proof of Concept, Open-Label Study Evaluating the Safety, Tolerability, and Efficacy of Regimens in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Safety, Tolerability, and Efficacy of Selonsertib, Firsocostat, and Cilofexor in Adults With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-384-3914
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — firsocostat

STUDY DESIGN:
Intervention Model Description: Cohorts 1-6 and 9 will be enrolled sequentially while Cohorts 7 and 8 will be randomized in parallel. Cohorts 10 and 11 will be randomized in parallel. Cohorts 12 and 13 will be randomized in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort 1: SEL 18 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive selonsertib (SEL) 18 mg tablet orally once daily for 12 weeks.
  Interventions: Drug: SEL
- Cohort 2: FIR 20 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive firsocostat (FIR) 20 mg tablet orally once daily for 12 weeks.
  Interventions: Drug: FIR
- Cohort 3: CILO 30 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive cilofexor (CILO) 30 mg tablet once daily for 12 weeks.
  Interventions: Drug: CILO
- Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive SEL 18 mg tablet + CILO 30 mg tablet once daily for 12 weeks.
  Interventions: Drug: SEL; Drug: CILO
- Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive SEL 18 mg tablet + FIR 20 mg tablet once daily for 12 weeks.
  Interventions: Drug: SEL; Drug: FIR
- Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive CILO 30 mg tablet + FIR 20 mg tablet once daily for 12 weeks.
  Interventions: Drug: FIR; Drug: CILO
- Cohort 7: CILO 20 mg (Cirrhotic) (Experimental): Participants with Child-Pugh-Turcotte Class A cirrhosis will receive FIR 20 mg tablet once daily for 12 weeks.
  Interventions: Drug: FIR
- Cohort 8: CILO 30 mg (Cirrhotic) (Experimental): Participants with Child-Pugh-Turcotte Class A cirrhosis will receive CILO 30 mg tablet once daily for 12 weeks.
  Interventions: Drug: CILO
- Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) (Experimental): Non-cirrhotic participants will receive SEL 18 mg tablet + FIR 20 mg tablet + CILO 30 mg tablet once daily for 12 weeks.
  Interventions: Drug: SEL; Drug: FIR; Drug: CILO
- Cohort 10: FIR 20 mg + FENO 48 mg (Experimental): Participants will receive fenofibrate (FENO) 48 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet + FENO 48 mg tablet orally once daily for 24 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH will be accepted to participate in this cohort.
  Interventions: Drug: FIR; Drug: FENO
- Cohort 11: FIR 20 mg + FENO 145 mg (Experimental): Participants will receive FENO 145 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet + FENO 145 mg tablet orally once daily for 24 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH will be accepted to participate in this cohort.
  Interventions: Drug: FIR; Drug: FENO
- Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g (Experimental): Participants will receive Vascepa® (VAS) 2 g capsule orally twice daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet once daily + CILO 30 mg tablet once daily + VAS 2 g capsule twice daily for 6 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH will be accepted to participate in this cohort.
  Interventions: Drug: FIR; Drug: CILO; Drug: VAS
- Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg (Experimental): Participants will receive FENO 145 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet once daily + CILO 30 mg tablet once daily + FENO 145 mg tablet orally once daily for 6 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH will be accepted to participate in this cohort.
  Interventions: Drug: FIR; Drug: CILO; Drug: FENO

INTERVENTIONS:
Drug: SEL — Administered orally once daily
  Other Names: GS-4997
  Arms: Cohort 1: SEL 18 mg (Non-cirrhotic); Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic); Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic); Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic)
Drug: FIR — Administered orally once daily
  Other Names: GS-0976
  Arms: Cohort 10: FIR 20 mg + FENO 48 mg; Cohort 11: FIR 20 mg + FENO 145 mg; Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g; Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg; Cohort 2: FIR 20 mg (Non-cirrhotic); Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic); Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic); Cohort 7: CILO 20 mg (Cirrhotic); Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic)
Drug: CILO — Administered orally once daily
  Other Names: GS-9674
  Arms: Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g; Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg; Cohort 3: CILO 30 mg (Non-cirrhotic); Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic); Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic); Cohort 8: CILO 30 mg (Cirrhotic); Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic)
Drug: FENO — Administered orally once daily
  Arms: Cohort 10: FIR 20 mg + FENO 48 mg; Cohort 11: FIR 20 mg + FENO 145 mg; Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Drug: VAS — Administered orally two times daily
  Arms: Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of selonsertib, firsocostat, cilofexor, fenofibrate and/or Vascepa® in adults with nonalcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females between 18-75 years of age (Cohorts 1-9: 18-75 years and Cohorts 10-13: ≥ 18 years); inclusive based on the date of the screening visit
* Willing and able to provide informed consent prior to any study specific procedures being performed
* For Cohorts 1 through 6 and 9, individuals must meet the following conditions:

  * Clinical diagnosis of nonalcoholic fatty liver disease (NAFLD)
  * Screening FibroTest® < 0.75, unless a historical liver biopsy within 12 months of Screening does not reveal cirrhosis. In individuals with Gilbert's syndrome or hemolysis, FibroTest® will be calculated using direct bilirubin instead of total bilirubin,
  * Screening magnetic resonance imaging - proton density fat fraction (MRI-PDFF) with ≥ 10% steatosis,
  * Screening magnetic resonance elastography (MRE) with liver stiffness ≥ 2.88 kPa, OR
  * A historical liver biopsy within 12 months of Screening consistent with NASH (defined as the presence of steatosis, inflammation, and ballooning) with stage 2-3 fibrosis according to the NASH Clinical Research Network (CRN) classification (or equivalent), AND
  * No documented weight loss > 5% between the date of the liver biopsy and Screening;
* For Cohorts 7 and 8, individuals must have a clinical diagnosis of NAFLD and have at least one of the following criteria:

  * Screening MRE with liver stiffness ≥ 4.67 kPa,
  * A historical FibroScan® ≥ 14 kPa within 6 months of Screening,
  * Screening FibroTest® ≥ 0.75,
  * A historical liver biopsy consistent with stage 4 fibrosis according to the NASH CRN classification (or equivalent);
* For Cohorts 10 and 11, individuals must have a clinical diagnosis of NAFLD and meet at least two criteria for metabolic syndrome modified from the NCEP ATP III Guidelines and one of the following criteria at Screening:

  * A historical liver biopsy within 6 months of Screening consistent with NASH and bridging fibrosis (F3) or within 12 months of Screening consistent with NASH and compensated cirrhosis (F4) in the opinion of the investigator,
  * Screening liver stiffness by MRE ≥ 3.64 kPa;
  * Screening liver stiffness by FibroScan® ≥ 9.9 kPa;
* For Cohorts 12 and 13, individuals must have a clinical diagnosis of NAFLD/NASH and at least two criteria for metabolic syndrome as modified from the NCEPT ATP III Guidelines, OR one of the following criteria:

  * A historical liver biopsy within 6 months of Screening consistent with NASH for individuals without compensated cirrhosis (F4); or within 12 months of Screening consistent with NASH for individuals with compensated cirrhosis (F4) in the opinion of the investigator,
  * A historical MRE with liver stiffness ≥ 2.88 kPa within 6 months of Screening,
  * A historical FibroScan® with liver stiffness ≥ 9.9 kPa within 6 months of Screening, AND
  * No documented weight loss > 5% between the date of the historical liver biopsy, historical MRE, or historical FibroScan® and Screening;
* Platelet count ≥ 100,000/µL;
* Serum creatinine < 2 mg/dL (Cohorts 1-9) at Screening;
* Estimated glomerular filtration rate (eGFR) ≥ 80 mL/min (Cohorts 10-11) or ≥ 60 mL/min (Cohorts 12-13), as calculated by the Cockcroft-Gault equation at Screening;
* For Cohorts 10-13, serum triglyceride level ≥ 150 mg/dL at Screening.

Key Exclusion Criteria:

* Pregnant or lactating females
* Other causes of liver disease including autoimmune, viral, and alcoholic liver disease
* Any history of decompensated liver disease, including ascites, hepatic encephalopathy or variceal bleeding
* For Cohorts 7-8, 10-13, Child-Pugh-Turcotte (CPT) score > 6
* History of liver transplantation
* History of hepatocellular carcinoma;
* Weight reduction surgery in the past 2 years or planned during the study;
* Documented weight loss > 5% between the date of the historical liver biopsy and Screening, if applicable;
* Body Mass Index (BMI) < 18 kg/m2;
* ALT > 5 x ULN at Screening;
* For Cohorts 10-13, HbA1c ≥ 9.5% (or serum fructosamine ≥ 381 µmol if HbA1c is unable to be resulted) at Screening;
* For Cohorts 10-13, hemoglobin ≤ 10.6 g/dL at Screening;
* INR > 1.2 (Cohorts 1-9) or INR > 1.4 (Cohorts 10-13) at Screening, unless on anticoagulation therapy;
* Total bilirubin > 1x ULN (Cohorts 1 through 6 and 9), >1.5 x ULN (Cohorts 7 and 8), or >1.3 x ULN (Cohorts 10-13) except in confirmed cases of Gilbert's syndrome;
* Triglycerides ≥ 500 mg/dL (Cohorts 5-8 and 10-13) or ≥ 250 mg/dL (Cohort 9) at Screening;
* Model for End-Stage Liver Disease (MELD) score > 12 at Screening (Cohorts 10 -13), unless due to an alternate etiology such as therapeutic anticoagulation;
* Chronic hepatitis B (HBsAg positive);
* Chronic hepatitis C (HCV RNA positive). individuals cured of HCV infection less than 2 years prior to the Screening visit are not eligible (Cohorts 10-13);
* HIV Ab positive;
* Presence of gallstones within 6 months of Screening (Cohorts 10-13);
* Alcohol consumption greater than 21 oz/week for males or 14 oz/week for females (1oz/30 mL of alcohol is present in 1 12oz/360 mL beer, 1 4oz/120 mL glass of wine, and a 1 oz/30 mL measure of 40% proof alcohol);
* Positive urine screen for amphetamines, cocaine or opiates (i.e., heroin, morphine) at Screening. Individuals on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to Screening may be included in the study. Individuals with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator;
* Unstable cardiovascular disease;
* History of intestinal resection of the extent that would result in malabsorption;
* Use of any prohibited concomitant medications as described in the protocol;
* History of a malignancy within 5 years of Screening with the following exceptions:

  * Adequately treated carcinoma in situ of the cervix,
  * Adequately treated basal or squamous cell cancer or other localized non-melanoma skin cancer.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (12):
  - Arizona Liver Health, Chandler, Arizona
  - Altman Clinical and Translational Research Clinic, La Jolla, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Hospital and Clinics (SHC), Stanford, California
  - Florida Research Institute, Lakewood Rch, Florida
  - Delta Research Partners, LLC, Bastrop, Louisiana
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Pinnacle Clinical Research, PLLC, Live Oak, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
- Auckland Clinical Studies Ltd, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawitz E, Neff G, Ruane P, Ziad Y, Jia C, Chuang J, et al. Fenofibrate Mitigates Increases in Serum Triglycerides Due to the ACC Inhibitor Firsocostat in Patients with Advanced Fibrosis Due to NASH. Poster presented at: The American Association for the Study of Liver Diseases (AASLD): The Liver Meeting; November 8-12, 2019; Boston, MA.
- [Background] Lawitz EJ, Coste A, Poordad F, Alkhouri N, Loo N, McColgan BJ, Tarrant JM, Nguyen T, Han L, Chung C, Ray AS, McHutchison JG, Subramanian GM, Myers RP, Middleton MS, Sirlin C, Loomba R, Nyangau E, Fitch M, Li K, Hellerstein M. Acetyl-CoA Carboxylase Inhibitor GS-0976 for 12 Weeks Reduces Hepatic De Novo Lipogenesis and Steatosis in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2018 Dec;16(12):1983-1991.e3. doi: 10.1016/j.cgh.2018.04.042. Epub 2018 Apr 26. PMID 29705265
- [Background] Lawitz E, Herring R, Younes ZH, Gane E, Ruane P, Schall RA, et al. Proof of Concept Study of an Apoptosis-Signal Regulating Kinase (ASK1) Inhibitor (Selonsertib) in Combination With An Acetyl-CoA Carboxylase Inhibitor (GS-0976) or a Farnesoid X Receptor Agonist (GS-9674) in Nash [Abstract PS-105]. European Association for the Study of the Liver (EASL); 2018 11-15 April; Paris, France.
- [Background] Lawitz E, Li K, Tarrant JM, Vimal M, Xu R, Song Q, et al. Hepatic de Novo Lipogenesis is Elevated in Patients with NASH Independent of Disease Severity [Abstract 2217]. American Association for the Study of Liver Diseases (AASLD); 2017 20-24 October Washington, DC.
- [Background] Lawitz EJ, Poordad F, Coste A, Loo N, Djedjos CS, McColgan B, et al. Acetyl-CoA carboxylase (ACC) inhibitor GS-0976 leads to suppression of hepatic de novo lipogenesis and significant improvements in MRI-PDFF, MRE, and markers of fibrosis after 12 weeks of therapy in patients with NASH [Abstract GS-009]. The International Liver Congress™ 2017: European Association for the Study of the Liver (EASL); 2017 19-23 April; Amsterdam, the Netherlands.
- [Result] Lawitz E, Bhandari BR, Ruane P, Kohli A, Harting E, Jia C, et al. Fenofibrate is Safe and Mitigates Increases in Serum Triglycerides in NASH Patients Treated with the Combination of the ACC Inhibitor Firsocostat and the FXR Agonist Cilofexor: A Randomized Trial. Poster presented at: The European Association for the Study of the Liver (EASL): International Liver Congress; June 23-26, 2021; Virtual Meeting.
- [Derived] Lawitz EJ, Bhandari BR, Ruane PJ, Kohli A, Harting E, Ding D, Chuang JC, Huss RS, Chung C, Myers RP, Loomba R. Fenofibrate Mitigates Hypertriglyceridemia in Nonalcoholic Steatohepatitis Patients Treated With Cilofexor/Firsocostat. Clin Gastroenterol Hepatol. 2023 Jan;21(1):143-152.e3. doi: 10.1016/j.cgh.2021.12.044. Epub 2022 Jan 6. PMID 34999207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in study sites in the United States and New Zealand. The first participant was screened on 13 June 2016. The last study visit occurred on 17 December 2020.
Groups:
- Cohort 1: SEL 18 mg (Non-cirrhotic): Non-cirrhotic participants received selonsertib (SEL) 18 mg tablet orally once daily for 12 weeks
- Cohort 2: FIR 20 mg (Non-cirrhotic): Non-cirrhotic participants received firsocostat (FIR) 20 mg tablet orally once daily for 12 weeks
- Cohort 3: CILO 30 mg (Non-cirrhotic): Non-cirrhotic participants received cilofexor (CILO) 30 mg tablet once daily for 12 weeks
- Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic): Non-cirrhotic participants received SEL 18 mg tablet + CILO 30 mg tablet once daily for 12 weeks
- Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic): Non-cirrhotic participants received SEL 18 mg tablet + FIR 20 mg tablet once daily for 12 weeks
- Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic): Non-cirrhotic participants received CILO 30 mg tablet + FIR 20 mg tablet once daily for 12 weeks
- Cohort 7: CILO 20 mg (Cirrhotic): Participants with Child-Pugh-Turcotte Class A cirrhosis received FIR 20 mg tablet once daily for 12 weeks
- Cohort 8: CILO 30 mg (Cirrhotic): Participants with Child-Pugh-Turcotte Class A cirrhosis received CILO 30 mg tablet once daily for 12 weeks
- Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic): Non-cirrhotic participants received SEL 18 mg tablet + FIR 20 mg tablet + CILO 30 mg tablet once daily for 12 weeks
- Cohort 10: FIR 20 mg + FENO 48 mg: Participants received FENO 48 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet + FENO 48 mg tablet orally once daily for 24 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
- Cohort 11: FIR 20 mg + FENO 145 mg: Participants received FENO 145 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet + FENO 145 mg tablet orally once daily for 24 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
- Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g: Participants received Vascepa® (VAS) 2 g capsule orally twice daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet once daily + CILO 30 mg tablet once daily + VAS 2 g capsule twice daily for 6 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
- Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg: Participants received FENO 145 mg tablet orally once daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet once daily + CILO 30 mg tablet once daily + FENO 145 mg tablet orally once daily for 6 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
Period: Pre-treatment Phase
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 16 | 33 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 16 | 30 | 32
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Investigator's Discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Phase
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Started | 10 (Only participants in Cohorts 10-13 received pre-treatment.) | 10 (Only participants in Cohorts 10-13 received pre-treatment.) | 10 (Only participants in Cohorts 10-13 received pre-treatment.) | 20 (Only participants in Cohorts 10-13 received pre-treatment.) | 20 (Only participants in Cohorts 10-13 received pre-treatment.) | 20 (Only participants in Cohorts 10-13 received pre-treatment.) | 10 (Only participants in Cohorts 10-13 received pre-treatment.) | 10 (Only participants in Cohorts 10-13 received pre-treatment.) | 13 (Only participants in Cohorts 10-13 received pre-treatment.) | 15 | 16 | 30 | 32
Completed | 10 | 10 | 10 | 20 | 20 | 19 | 10 | 9 | 13 | 15 | 15 | 28 | 32
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: SEL 18 mg (Non-cirrhotic): Non-cirrhotic participants received SEL 18 mg tablet orally once daily for 12 weeks
- Cohort 2: FIR 20 mg (Non-cirrhotic): Non-cirrhotic participants received FIR 20 mg tablet orally once daily for 12 weeks
- Cohort 3: CILO 30 mg (Non-cirrhotic): Non-cirrhotic participants received CILO 30 mg tablet once daily for 12 weeks
- Cohort 10: FIR 20 mg + FENO 48 mg: Participants received FENO 48 mg tablet orally for 2 weeks in the pretreatment phase, then FIR 20 mg tablet + FENO 48 mg tablet orally once daily for 24 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
- Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g: Participants received VAS 2 g capsule orally twice daily for 2 weeks in the pretreatment phase, then FIR 20 mg tablet once daily + CILO 30 mg tablet once daily + VAS 2 g capsule twice daily for 6 weeks in the treatment phase. Participants with compensated cirrhosis due to NASH were accepted to participate in this cohort.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 20 | 20 | 10 | 10 | 13 | 15 | 16 | 30 | 32 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.0) | 57 (9.8) | 53 (12.3) | 56 (7.8) | 48 (13.8) | 55 (10.7) | 60 (11.1) | 60 (9.5) | 56 (8.2) | 59 (9.7) | 52 (14.2) | 56 (11.1) | 52 (11.5) | 55 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 9 | 13 | 11 | 12 | 7 | 6 | 11 | 10 | 9 | 24 | 22 | 148
  Male | 1 | 5 | 1 | 7 | 9 | 8 | 3 | 4 | 2 | 5 | 7 | 6 | 10 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 8 | 12 | 5 | 11 | 6 | 3 | 9 | 2 | 10 | 15 | 17 | 115
  Not Hispanic or Latino | 2 | 1 | 2 | 8 | 15 | 9 | 4 | 7 | 4 | 13 | 6 | 15 | 15 | 101
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 10 | 10 | 10 | 19 | 17 | 17 | 10 | 10 | 12 | 14 | 16 | 30 | 30 | 205
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7
  United States | 10 | 10 | 10 | 20 | 17 | 17 | 10 | 10 | 12 | 15 | 16 | 30 | 32 | 209

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events
Description: Treatment-emergent AEs were defined as events that met 1 or both of the following criteria:
  * Any AEs with onset dates on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
  * Any AEs leading to premature discontinuation of study drug
Time Frame: Cohorts 1-9: First dose date up to 12 weeks plus 30 days; Cohorts 10-11: First dose date up to 26 weeks plus 30 days; Cohorts 12-13: First dose date up to 8 weeks plus 30 days. For Cohorts 10-13, the first dose date included the Pre-treatment Phase.
Population: The Safety Analysis Set included all participants who were administered at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 20 | 20 | 10 | 10 | 13 | 15 | 16 | 30 | 32
percentage of participants | 50 | 60 | 50 | 25 | 40 | 50 | 80 | 70 | 76.92 | 86.67 | 87.5 | 40 | 37.5

2. Primary Outcome: Percentage of Participants Who Experienced Treatment Emergent Serious Adverse Events
Description: A treatment emergent serious adverse event (SAE) was defined as an event that, at any dose, results in the following:
  * Death
  * Life-threatening
  * In-patient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * A congenital anomaly/birth defect
  * A medically important event or reaction
Time Frame: as for outcome 1
Population: The Safety Analysis Set included all participants who were administered at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 20 | 20 | 10 | 10 | 13 | 15 | 16 | 30 | 32
percentage of participants | 0 | 0 | 0 | 5 | 5 | 5 | 10 | 0 | 7.69 | 0 | 0 | 3.33 | 3.12

3. Primary Outcome: Percentage of Participants Who Experienced Grade 3 or Higher Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug. If baseline laboratory data were missing, then any abnormality of at least Grade 1 was considered treatment emergent. Graded laboratory abnormalities were defined using the grading scheme in the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 for Cohorts 1-9 and CTCAE Version 5.0 for Cohorts 10-13.
Time Frame: as for outcome 1
Population: The Safety Analysis Set included all participants who were administered at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 20 | 20 | 10 | 10 | 13 | 15 | 16 | 30 | 32
percentage of participants | 20 | 20 | 40 | 10 | 20 | 10 | 40 | 30 | 15.4 | 6.7 | 12.5 | 6.7 | 6.3

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose (Cohorts 1-9: up to 12 weeks; Cohorts 10-11: up to 26 weeks; Cohorts 12-13: up to 8 weeks) plus 30 days. For Cohorts 10-13, the first dose date included the Pre-treatment Phase. All-cause Mortality: Cohorts 1 through 6 and 9: Enrollment up to 12 weeks plus 30 days; Cohorts 7-8: Randomization up to 12 weeks plus 30 days; Cohorts 10-11: Randomization up to 26 weeks plus 30 days; Cohort 12-13: Randomization up to 8 weeks plus 30 days
Description: Adverse Events: The Safety Analysis Set included all participants who were administered at least 1 dose of the study drug.
  All-cause Mortality: All Enrolled Analysis Set included all participants in Cohorts 1 through 6 and 9 who received a study subject identification number in the study after screening. The Randomized Analysis Set included all participants who were randomized into Cohorts 7, 8, and Cohorts 10-13.
Arm/Group | Cohort 1: SEL 18 mg (Non-cirrhotic) | Cohort 2: FIR 20 mg (Non-cirrhotic) | Cohort 3: CILO 30 mg (Non-cirrhotic) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) | Cohort 7: CILO 20 mg (Cirrhotic) | Cohort 8: CILO 30 mg (Cirrhotic) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) | Cohort 10: FIR 20 mg + FENO 48 mg | Cohort 11: FIR 20 mg + FENO 145 mg | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/20 | 0/20 | 0/20 | 0/10 | 0/10 | 0/13 | 0/15 | 0/16 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/20 | 1/20 | 1/20 | 1/10 | 0/10 | 1/13 | 0/15 | 0/16 | 1/30 | 1/32
Other Adverse Events (participants affected / at risk) | 5/10 | 6/10 | 5/10 | 5/20 | 8/20 | 10/20 | 8/10 | 7/10 | 10/13 | 13/15 | 14/16 | 7/30 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SEL 18 mg (Non-cirrhotic) (N=10) | Cohort 2: FIR 20 mg (Non-cirrhotic) (N=10) | Cohort 3: CILO 30 mg (Non-cirrhotic) (N=10) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) (N=20) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) (N=20) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) (N=20) | Cohort 7: CILO 20 mg (Cirrhotic) (N=10) | Cohort 8: CILO 30 mg (Cirrhotic) (N=10) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) (N=13) | Cohort 10: FIR 20 mg + FENO 48 mg (N=15) | Cohort 11: FIR 20 mg + FENO 145 mg (N=16) | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g (N=30) | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg (N=32)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SEL 18 mg (Non-cirrhotic) (N=10) | Cohort 2: FIR 20 mg (Non-cirrhotic) (N=10) | Cohort 3: CILO 30 mg (Non-cirrhotic) (N=10) | Cohort 4: SEL 18 mg + CILO 30 mg (Non-cirrhotic) (N=20) | Cohort 5: SEL 18 mg + FIR 20 mg (Non-cirrhotic) (N=20) | Cohort 6: CILO 30 mg + FIR 20 mg (Non-cirrhotic) (N=20) | Cohort 7: CILO 20 mg (Cirrhotic) (N=10) | Cohort 8: CILO 30 mg (Cirrhotic) (N=10) | Cohort 9: SEL 18 mg + FIR 20 mg + CILO 30 mg (Non-cirrhotic) (N=13) | Cohort 10: FIR 20 mg + FENO 48 mg (N=15) | Cohort 11: FIR 20 mg + FENO 145 mg (N=16) | Cohort 12: FIR 20 mg + CILO 30 mg + VAS 2g (N=30) | Cohort 13: FIR 20 mg + CILO 30 mg + FENO 145 mg (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 2 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 5 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 5 | 1 | 4 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal atrophy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met.

* The results of the study in their entirely have been publicly disclosed by our with the consent of Gilead in an abstract, manuscript, presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02781584/Prot_000.pdf
  • Statistical Analysis Plan: Cohort 1-9 SAP (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02781584/SAP_001.pdf
  • Statistical Analysis Plan: Cohort 10-11 SAP (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02781584/SAP_002.pdf
  • Statistical Analysis Plan: Cohort 12-13 SAP (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02781584/SAP_003.pdf